CLINICAL TRIAL: NCT00547651
Title: AMR PH GL 2007 CL001 Phase 3 A Randomized, Open-Label, Multinational Phase 3 Trial Comparing Amrubicin Versus Topotecan in Patients With Extensive or Limited and Sensitive or Refractory Small Cell Lung Cancer After Failure of First-Line Chemotherapy
Brief Title: AMR PH GL 2007 CL001 Phase 3 Trial in Patients With Small Cell Lung Cancer After Failure of First-Line Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMR PH GL 2007 CL001
Record Dates: First submitted 2007-10-18; First posted 2007-10-22 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-10

CONDITIONS: Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; Lung Cancer; Limited Disease Sensitive Small Cell Lung Cancer; Extensive Disease Sensitive Small Cell Lung Cancer; Limited Disease Refractory Small Cell Lung Cancer; Extensive Disease Refractory Small Cell Lung Cancer; Refractory Small Cell Lung Cancer; Sensitive Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — amrubicin; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amrubicin (Experimental): Amrubicin
  Interventions: Drug: Amrubicin
- Topotecan (Active Comparator): Topotecan
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: Amrubicin — Amrubicin for injection is supplied as 50-mg vials. Patients will receive 40 mg/m2 amrubicin as a 5-minute infusion once daily for 3 consecutive days starting on Day 1 of a 21-day course
  Other Names: amrubidin hydrochloride; Calsed; CNF3140
  Arms: Amrubicin
Drug: Topotecan — Topotecan for injection is supplied as 4-mg vials. Patients will receive 1.5 mg/m2 as a 30-minute infusion once daily for 5 consecutive days starting on Day 1 of a 21-day course
  Other Names: Topotecan hydrochloride; Hycamtin
  Arms: Topotecan

SUMMARY:
This study drug (Amrubicin) is believed to work by stopping the tumor cells in your body from growing. The purpose of this study is to evaluate the effect of amrubicin compared to topotecan in the treatment of small cell lung cancer.

DETAILED DESCRIPTION:
Small cell lung cancer represents approximately 13% of the cancers of the lung and presents as extensive stage disease in 60% to 70% of patients. Sites of metastases include bone (35%), liver (25%), bone marrow (20%), brain (10%), extrathoracic lymph nodes (5%), and subcutaneous masses (5%). Small-cell lung cancer has prominent markers of neuroendocrine differentiation.

The staging classification for SCLC is the 2-stage Veterans Administration Lung Study Group system that categorizes patients as having limited or extensive disease. Limited stage SCLC is disease confined to 1 hemithorax with or without adjacent mediastinal and/or supraclavicular lymph node involvement, but without a pleural effusion. This extent of disease can be included in a tolerable radiation field. Extensive-disease SCLC is any disease beyond the definition of limited-stage disease.

There are few proven treatment options for SCLC patients who fail first-line chemotherapy. New treatment strategies must be evaluated. The need to discover active agents with better toxicity profiles continues to be of great importance. Amrubicin may be an effective treatment for this population.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of SCLC at study entry according to the International Association for the Study of Lung Cancer (IASLC) histopathologic classification. Mixed or combined subtypes according to the IASLC are not allowed;
* SCLC that is either sensitive (defined as a response including stable disease to first-line platinum-based chemotherapy, with subsequent progression >/= 90 days after completing first-line chemotherapy) or refractory (defined as best response to first-line platinum-based chemotherapy or progression < 90 days after completing first-line chemotherapy);
* Extensive or limited disease; patients with limited disease who are candidates for local or regional salvage radiation therapy must have been offered such treatment prior to participation in this study;
* Radiographically documented progression after first-line treatment with platinum-based chemotherapy;
* No more than 1 prior chemotherapy regimen;
* At least 18 years of age;
* ECOG performance status of 0 - 1

Exclusion Criteria:

* Chest radiotherapy with curative intent to the primary disease complex </= 28 days prior to first dose; CNS radiotherapy </= 21 days prior to first dose; radiotherapy to all other areas </= 7 days prior to first dose;
* Prior anthracycline, topotecan, or irinotecan treatment.
* Prior anthracycline or topotecan treatment.
* Patients with know history of seropositive human immunodeficiency virus (HIV) or patients who are receiving immunosuppressive medications that would increase the risk of serious neutropenic complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 637 (Actual)
Dates: Start 2007-09-01 (Actual); Primary Completion 2011-05-01 (Actual); Study Completion 2011-05-01 (Actual)

PRIMARY OUTCOMES:
The primary objective is to demonstrate superiority in overall survival of amrubicin compared with topotecan hydrochloride in patients with small cell lung cancer (SCLC) after failure of first-line chemotherapy. | Until death from any cause

SECONDARY OUTCOMES:
To further characterize the clinical benefit of amrubicin compared with topotecan in terms of objective response rate | Until death
To further characterize the clinical benefit of amrubicin compared with topotecan in terms of progression-free survival. | Until death
To further characterize the clinical benefit of amrubicin compared with topotecan in terms of duration of response | Until death
To further characterize the clinical benefit of amrubicin compared with topotecan in terms of time to tumor progression | Until death
To further characterize the clinical benefit of amrubicin compared with topotecan in terms of safety | Until death
To further characterize the clinical benefit of amrubicin compared with topotecan in terms of quality of life | Until death

CONTACTS AND LOCATIONS:
Overall Officials: Markus Renschler, M.D., Study Director — Celgene Corporation
Locations (140):
- United States (61):
  - Northwest Alabama Cancer Center, Muscle Shoals, Alabama
  - Arizona Oncology Associates, Tucson, Arizona
  - Little Rock Hematology Oncology Associates, Little Rock, Arkansas
  - Cancer Care Associates of Fresno Medical Group, Inc., Fresno, California
  - Cedars-Sinai Outpatient Cancer Center, Los Angeles, California
  - University of Colorado Health Science Centre, Aurora, Colorado
  - Rocky Mountain Cancer Center - Midtown (Main), Denver, Colorado
  - Advanced Medical Specialties, Miami, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Centers of Florida, P.A., Ocoee, Florida
  - Florida Oncology Associates, Orange Park, Florida
  - Sacred Heart Medical Oncology, Pensacola, Florida
  - Medical Oncology Associates of Augusta, Augusta, Georgia
  - Joliet Oncology-Hematology Associates, Ltd., Joliet, Illinois
  - Cancer & Hematology Specialists of Chicago (Main), Niles, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Cancer Care at Blessing Hospital, Quincy, Illinois
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Hope Center, Terre Haute, Indiana
  - Kansas City Cancer Center (Main), Overland Park, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Jayne Gurtler MD, Laura Brizn MD, Angelo Russo MD, and Janet Burroff MD, APMC, Metairie, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Maine Center for Cancer Medicine and Blood Disorders, Scarborough, Maine
  - Sinai Hospital of Baltimore, Inc., Baltimore, Maryland
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Alliance Hematology Oncology, P.A. (Main), Westminster, Maryland
  - Kalamazoo Hematology and Oncology, Kalamazoo, Michigan
  - Michigan Hematology & Oncology Institute, Southgate, Michigan
  - University of Minnesota Medical Center, Cancer Center, Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - St. Joseph Oncology, Inc., Saint Joseph, Missouri
  - Comprehensive Care Centers of Nevada (Main), Las Vegas, Nevada
  - New York Oncology Hematology, P.C., Latham, New York
  - SUNY Upstate Medical University - Regional Oncology Center, Syracuse, New York
  - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Regional Cancer Care, Durham, North Carolina
  - Cancer Centers of North Carolina (Main), Raleigh, North Carolina
  - Piedmont Hematology Oncology Associates, Winston-Salem, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Greater Dayton Cancer Center (Main), Kettering, Ohio
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Cancer Care Associates, Tulsa, Oklahoma
  - Willamette Valley Cancer Center (Main), Eugene, Oregon
  - Medical Oncology Associates, Kingston, Pennsylvania
  - Thomas Jefferson Memorial Hospital, Philadelphia, Pennsylvania
  - UPMC Cancer Pavilion, Pittsburgh, Pennsylvania
  - Cancer Centers of the Carolinas (Main), Greenville, South Carolina
  - The Sarah Cannon Research Institute/TN Oncology, Nashville, Tennessee
  - Texas Oncology, P.A., Amarillo, Texas
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - Texas Cancer Center at Medical City (Main), Dallas, Texas
  - Texas Oncology, P.A. (Main), Dallas, Texas
  - West Texas Cancer Center-Texas Oncology, Odessa, Texas
  - Texas Oncology, P.A., Webster, Texas
  - Texoma Cancer Center, Wichita Falls, Texas
  - Fairfax Northern Virginia Hematology/Oncology, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - Northwest Cancer Specialists - Vancouver (Main), Vancouver, Washington
  - Marshfield Clinic, Marshfield, Wisconsin
- Australia (5):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - New South Wales Southern Medical Day Care Centre, Wollongong, New South Wales
  - The Princess Alexandra Hospital, Dept of Respiratory Medicine, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Queen Elizabeth Hospital, Woodville South
- Austria (4):
  - Allgemeines Krankenhaus der Stadt Linz, Abteilung fur Atem und Lungenkrankheiten, Linz
  - Allegemeines Krankenhaus Wien, Univ. Klinik fur Innere, Medizin I, Vienna
  - Krankenhaus Hietzing, 5 Med. Abteilung mit Onkologie, Vienna
  - Klinikum Weis-Grieskirchen GmbH, Wels
- Belgium (5):
  - UZ Brussel, Medical Oncology and Hematology, Brussels
  - Centre Hospitalier Notre-Dame et Reine Fabiola, Charleroi
  - Universitair Ziekenhuis Antwerpen, Dept. Respiratory Diseases, Edegem
  - UZ Gasthuisberg, UZ Leuven, Leuven
  - C.H.U. Sart-Tilman, Liège
- Bulgaria (4):
  - III-rd Internal Department, District Dispensary for Oncology diseases with stationary(DDOncDIU), Plovdiv
  - DDOncDIU Sofia District, Sofia
  - MHAT "Tsaritsa Yoanna", Sofia
  - University Multiprofile Hospital for Active Treatment "Sveta Marina", Varna
- Canada (5):
  - Fraser Valley Cancer Centre-Surrey Memorial Hospital, Surrey, British Columbia
  - London Regional Cancer Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Humber River Regional Hospital, Weston, Ontario
  - Royal Victoria Hospital, Montreal, Quebec
- Czechia (4):
  - Fakultni Nemocnice Ostrava, Ostrava-Poruba
  - Fakultní Thomayerova nemocnice s poliklinikou, Prague
  - Faculty Hospital Motol, Prague
  - Masarykova nemocnice v Ústí nad Labem, Ústí nad Labem
- Denmark (3):
  - Rikshospitalet, Finsen Center, Copenhagen
  - Herlev Hospital, Onkologisk afdeling R, Herlev
  - Odense Universitetshospital,Onkologisk afdeling R, Odense C
- France (4):
  - Centre François Baclesse, Caen
  - Hôpital de la Croix-Rousse, Lyon
  - CHU Montpellier - Unité de Cancérologie Thoracique, Montpellier
  - Institut Gustave Roussy, Villejuif
- Germany (10):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Charité Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Essen Innere Klinik und Poliklinik, Essen
  - Asklepios Fachkliniken Muenchen Gauting, Gauting
  - Krankenhaus Grosshansdorf, Zentrum fur Pneumologie und Thoraxchirurgie, Großhansdorf
  - Staedtisches Krankenhaus Martha-Maria Halle-Doelau, Halle
  - Thoraxklinik am Universitätsklinikum Heidelberg AG, Heidelberg
  - St. Vincentius-Kliniken Karlsruhe, Hamatologie, Med Onkologie und Immunologie, Karlsruhe
  - Katholisches Klinikum Mainz, St. Hildegardis Krankenhaus, Mainz
  - Klinikum Mannheim GmbH, Chirugische Klinik, Thorakale Onkologie, Mannheim
- Hungary (6):
  - Semmelweis University of Medicine, Budapest
  - Országos Korányi Tbc és Pulmonológiai Intézet, Budapest
  - DEODEC, Debrecen
  - Matrai Gyogyintezet, Mátraháza
  - County Hospital Baranya, Pécs
  - Erzsébet Hospital Sopron, Sopron
- Italy (4):
  - Policlinico di Modena - University of Modena & Reggio Emilia, Dept Oncology & Hematology, Modena
  - Ospedale S. Maria della Misericordia, Perugia
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Ospedale S.S. Trinita, Sora
- Netherlands (5):
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - VU University Medical Center Amsterdam, Amsterdam
  - University Medical Center Groningen, Groningen
  - Elkerliek Ziekenhuis, Locatie Helmond, Helmond
  - Erasmus MC - Daniel den Hoed, Rotterdam
- Poland (8):
  - Specjalistyczny Zespol Chorob Pluc i Gruzlicy w Bystrej, Bystra
  - Akademickie Centrum Kliniczne, Gdansk
  - Zespol nr 1 Szpitala im. St. Leszczynskiego, Katowice
  - Klinika Nowotworow Ukladowych i Uogolnionych Centrum Onkologii, Instytut im. Marii Sklodowskiej-Curie, Krakow
  - Centrum Onkologii Ziemi Lubelskiej, Lublin
  - Wielkopolskie Centrum Pulmonologii i Tarakochirurgii Oddzial Onkologii Klinicznej z Pododdzialem Dziennej Chemioterapii, Poznan
  - Szpital Specjalistyczny w Prabutach, Prabuty
  - Wojewódzki Szpital Chorób Pluc im Alojzego Pawelca w Wodzislawiu Slaskim, Wodzisław Śląski
- Spain (5):
  - Hospital Universitario Germans Trias i Pujol, Barcelona
  - Duran i Reynals Institut Catala d'Oncologia, L'Hospitalet de Llobregat
  - Fundación Jiménez Díaz. Universidad Autónoma de Madrid, Madrid
  - Hospital Universitario Virgin de la Victoria, Málaga
  - Hospital General Universitario de Valencia, Valencia
- Switzerland (3):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Graubünden, Chur
  - Universitätsspital Zürich, Zurich
- United Kingdom (4):
  - Edinburgh Cancer Research Centre, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Christie Hospital NHS Foundation Trust, Manchester
  - The Royal Marsden NHS Foundation Trust, Surrey

REFERENCES:
- [Background] von Pawel J, Jotte R, Spigel DR, O'Brien ME, Socinski MA, Mezger J, Steins M, Bosquee L, Bubis J, Nackaerts K, Trigo JM, Clingan P, Schutte W, Lorigan P, Reck M, Domine M, Shepherd FA, Li S, Renschler MF. Randomized phase III trial of amrubicin versus topotecan as second-line treatment for patients with small-cell lung cancer. J Clin Oncol. 2014 Dec 10;32(35):4012-9. doi: 10.1200/JCO.2013.54.5392. Epub 2014 Nov 10. PMID 25385727